CLINICAL TRIAL: NCT07219199
Title: Intraoperative Quantification of Residual IDH1-mutant Tumor Cells Via Ultra-Rapid Droplet Digital PCR
Brief Title: Residual IDH1-Mutant Tumor Cell Quantification Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pending-IDE G250266
Record Dates: First submitted 2025-10-20; First posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- UR-ddPCR During Tumor Biopsy/Resection Procedure (Experimental): During the participant's tumor biopsy or resection, the neurosurgeon will perform maximal safe resection, as per standard clinical practice, and allocate nine tissue specimens (three from the core of the tumor and six from the tumor-brain interface) for UR-ddPCR testing. If both core and tumor-brain interface samples test positive and further removal is judged safe, the neurosurgeon may perform additional resection and obtain final specimens from the positive sites before concluding the surgery. Up to 15 tissue specimens may be collected and tested during the procedure. Postoperative care and clinical follow-up will proceed per standard of care.
  Interventions: Device: UR-ddPCR

INTERVENTIONS:
Device: UR-ddPCR — The investigational UR-ddPCR assay will be performed on collected tissue specimens during the participant's scheduled surgical visit.

SUMMARY:
This is a single-site, single-arm, prospective, interventional cohort study using intraoperative ultra-rapid droplet digital polymerase chain reaction (UR- ddPCR) to assess residual IDH1-mutant tumor at the end of surgical resection and, if positive, guide additional resection in real-time.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of consent (any sex)
* Newly diagnosed diffuse glioma with either (a) radiographic features consistent with IDH-mutant glioma or (b) prior molecular confirmation of an IDH mutation
* Scheduled for tumor tissue biopsy or surgical resection at NYU Langone Health

Exclusion Criteria:

• Active hepatitis C virus (HCV) infection or suspected/confirmed prion disease (e.g., Creutzfeldt-Jakob disease), as documented in the medical record or by the treating physician, due to biosafety and tissue- handling restrictions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to Year 3 Post-Procedure
  PFS is defined as the time from surgery to the time of the first MRI demonstrating radiographic progression (using Response Assessment in Neuro-Oncology [RANO] criteria) or death due to any cause (whichever occurs earlier).

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to Year 3 Post-Procedure
  OS is defined as the time from surgery to the time of death due to any cause (whichever occurs earlier).
Residual Tumor Volume | Postoperative Day 1 (POD1)
  Assessed via MRI.
Radiographic PFS | Month 6 Post-Procedure, Month 12 Post-Procedure, Month 24 Post-Procedure, Month 36 Post-Procedure
  Radiographic PFS is defined as the time from surgery to the time of the first MRI demonstrating radiographic progression (using Response Assessment in Neuro-Oncology [RANO] criteria).
Time to Radiographic Recurrence | Up to Year 3 Post-Procedure
  Time to Radiographic Recurrence is defined as the time from surgery to the time of the first MRI demonstrating radiographic recurrence.
Percent Change in Mutant Allele Fraction (MAF) | Post-Operative Day 0 (POD0), post-additional resection of tumor-brain interface samples (Up to Year 3)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Orringer, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided